CLINICAL TRIAL: NCT05594849
Title: Evaluation of Efficacy, Safety and Patient' Satisfaction of Therapeutic Switch From Off-Label Swallowed Steroids to Budesonide Orodispersible Tablets (Jorveza) in Eosinophilic Esophagitis: a Prospective Observational Study
Brief Title: Evaluation of Efficacy, Safety and Patient' Satisfaction of Therapeutic Switch From Off-Steroids to Budesonide
Acronym: Switch
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2711
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Budesonide Orodispersible Tablets (Jorveza) — Patients that swith to Budesonide Orodispersible Tablets (Jorveza)

SUMMARY:
Eosinophilic esophagitis (EoE) is a chronic, immune-mediated, esophageal-restricted disease characterized clinically by symptoms related to esophageal dysfunction and histologically by an eosinophil-predominant inflammation.A dramatic increase in incidence and prevalence of EoE has been documented over the last 2 decades, especially in Western countries.EoE is currently the most common cause of dysphagia and bolus impaction, and the second leading cause of chronic esophagitis after gastroesophageal reflux disease.Predominant symptoms of EoE in adult patients are chronic dysphagia, food impaction, and chest pain.EoE is a chronic-progressive disease and, if left untreated, is usually associated with persistence of symptoms and inflammation.Furthermore, it is well established that the ongoing eosinophilic inflammation leads to esophageal remodeling, resulting in fibrosis with possible stricture formation and functional damage.Consequently, EoE has a substantial negative impact on the health-related quality of life (HRQoL) of patients and their families by causing emotional distress and restricting social activities.There is, therefore, a clear indication to treat patients suffering from active EoE.

Today, swallowed topical-acting corticosteroids (STCs) are an established first-line pharmacologic treatment for patients with EoE.Proton pump inhibitors (PPIs) and dietary modifications are alternatives. From the first positive attempt to treat EoE with STCs, drugs that were originally developed for airway administration in patients with asthma and used off-label in eosinophilic esophagitis,multiple trials have confirmed the efficacy of these compounds in improving symptoms as well as inflammation in patients with EoE. Fluticasone or budesonide have shown comparable potencies, but the vehicle depositing the compound on the esophageal surface seems to be critical.Until now there has been no licensed therapy for eosinophilic esophagitis treatment; treatment using drugs adapted from other conditions has been limited and not standardized.

Recently a new budesonide orodispersible tablet formulation (BOT, originally defined as an "effervescent tablet for orodispersible use [BET]") has been created and has been shown in clinical trials to be able to resolve both the symptoms and the underlying inflammation in EoE in most patients.

Budesonide orodispersible tablet treatment has been shown to be significantly more effective than placebo in inducing clinical and histologic remission in patients affected by EoE. A phase 3 trial showed the effectiveness of a 6-week treatment with new budesonide orodispersible tablet (BOT) to induce clinicohistologic remission in 58% of adult patients with EoE, which increased to 85% when therapy was extended to 12 weeks in nonresponders.

Another clinical trial showed that after 48 weeks of treatment, 73.5% of patients treated with low-dose and 75% of patients treated with high dose budesonide remained in remission, compared with 4.4% of patients treated with placebo.

The budesonide orodispersible tablet formulation, with the name of Jorveza, received the marketing authorization valid in the EU on 8 January 2018 and recently received AIFA approval to be distributed in Italy as the first medicine with indication for eosinophilic esophagitis.

Therefore, patients with eosinophilic esophagitis who are taking off-label corticosteroid formulations (fluticasone diproprionate and budesonide in galenic formulation) will need to make a therapeutic transition to Jorveza.

No data are currently available in the literature about efficacy, safety and patient' satisfaction after therapeutic switch from off-label swallowed topical-acting corticosteroids to budesonide orodispersible tablet formulation (Jorveza).

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of eosinophilic esophagitis (> 15 eosinophils / HPF in at least one esophageal biopsy and symptoms of esophageal dysfunction)
* therapy with off-label topical steroid therapy (fluticasone or budesonide) within the last 3 months
* availability of EGDS + histological results performed during off-label topical steroid therapy in the last 6 months
* Signed informed consent form

Exclusion Criteria:

* age <16 or> 80 years
* intolerance to Jorveza or to any of the excipients
* arbitrary suspension of treatment during the study period

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment | 12 months
  Number of AE/SAE of patients, number of patients with endoscopic remission of the disease, tolerability and appreciation of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No